CLINICAL TRIAL: NCT05645159
Title: Effectiveness of a Heart Disease Blended Learning Program in Future Physiotherapy Professionals: A Prospective Study
Brief Title: Blended Learning in Future Physiotherapy Professionals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, David Hernández-Guillén, Assistant professor, PT, PhD, University of Valencia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BL_HEART_01
Record Dates: First submitted 2022-11-25; First posted 2022-12-09 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Heart Diseases; Teach-Back Communication
Keywords: Blended learning; Education; Teaching methods; Physiotherapy; Students
MeSH Terms: conditions — Heart Diseases; Teach-Back Communication

STUDY DESIGN:
Intervention Model Description: Students of physiotherapy of the University of Valencia
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Physiotherapy students (Experimental): The participants performed an 8-week heart disease blended learning program.
  Interventions: Other: Blended learning in heart disease

INTERVENTIONS:
Other: Blended learning in heart disease — The intervention included face-to-face classes and online resources (Moodle, online syllabus, videos, websites, podcasts, activities, apps, forums, emails, tutoring).

SUMMARY:
Blended Learning (BL) is proving to be an effective method of teaching within the health professions . However, there are still scarce studies on BL conducted with undergraduate physiotherapy students. Therefore, the aim of this study was to determine the effectiveness of a heart disease BL programme in knowledge, motivation, engagement, design of the programme instructions and learning behaviours in physiotherapy students.

ELIGIBILITY:
Inclusion Criteria:

* studying a Physiotherapy Degree at the aforementioned University
* to be willing to participate

Exclusion Criteria:

* none

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 124 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Coronary Artery Disease Education Questionnaire (CADEQ) | 0 weeks
  CADEQ includes 20 closed-ended questions about medical conditions, risk factors, exercise, nutrition, and psychosocial wellbeing with a single-word answer (yes, no). Total score ranges from 0 to 20 (0=poorest knowledge, 20=best knowledge).
Coronary Artery Disease Education Questionnaire (CADEQ) | 4 weeks
  CADEQ includes 20 closed-ended questions about medical conditions, risk factors, exercise, nutrition, and psychosocial wellbeing with a single-word answer (yes, no). Total score ranges from 0 to 20 (0=poorest knowledge, 20=best knowledge).
Coronary Artery Disease Education Questionnaire (CADEQ) | 8 weeks
  CADEQ includes 20 closed-ended questions about medical conditions, risk factors, exercise, nutrition, and psychosocial wellbeing with a single-word answer (yes, no). Total score ranges from 0 to 20 (0=poorest knowledge, 20=best knowledge).
Coronary Artery Disease Education Questionnaire (CADEQ) | 12 weeks
  CADEQ includes 20 closed-ended questions about medical conditions, risk factors, exercise, nutrition, and psychosocial wellbeing with a single-word answer (yes, no). Total score ranges from 0 to 20 (0=poorest knowledge, 20=best knowledge).
Coronary Artery Disease Education Questionnaire (CADEQ) | 20 weeks
  CADEQ includes 20 closed-ended questions about medical conditions, risk factors, exercise, nutrition, and psychosocial wellbeing with a single-word answer (yes, no). Total score ranges from 0 to 20 (0=poorest knowledge, 20=best knowledge).

SECONDARY OUTCOMES:
Effect of the Dader Method in Cardiovascular Risk of Patients with Risk Factors or Cardiovascular Disease Questionnaire (EMDADER) | 0, 4, 8, 12 and 20 weeks
  EMDADER is composed of 10 multiple-choice questions with four answer options on coronary artery disease and risk factors, and two questions to report weight and height. Total score ranges from 0 to 10 (0=poorest knowledge, 10=best knowledge).
Academic Motivation Scale and Attributional Styles Questionnaire | 4, 8 weeks
  The tool is composed of 24 items, using a 7-point Likert scale: from 1 (totally disagree) to 7 (totally agree). The scale integrates three domains related to learning motivation: Intrinsic Motivation (9 items), Performance Motivation (7 items) and Extrinsic Motivation (7 items). The maximum score is 7. The scale is prepared to add the different items even if they measure different items. They will not be interpreted separately.
Student Engagement Questionnaire | 4, 8 weeks
  It is a 35-item questionnaire, scored on a five-point Likert scale (1=totally disagree, 5=totally agree). The questionnaire is divided into five dimensions: Intellectual Capabilities (items 1-10), Working Together (items 11-16), Teaching (items 17-25), Teacher-student Relationship (items 26-29), and Student-student Relationship (items 30-35). The maximum score of the questionnaire is 5. The scale is prepared to add the different items even if they measure different items. They will not be interpreted separately.
Community of Inquiry Survey | 0, 4, 8, 12 and 20 weeks
  A 34-item questionnaire, scored on a five-point Likert scale (1=strongly disagree, 5=strongly agree) that includes three dimensions: i) Cognitive Presence (items 1-13), related to the degree to which participants are able to construct meaning and knowledge through continuous communication, reflection, and discussion; ii) Social Presence (items 14-22), related to the ability of participants to identify with the community, communicating and developing interpersonal relationships; iii) Teaching Presence (items 23-34), referring to the design, guidance and direction, on the part of teachers, of cognitive and social processes with the purpose of achieving the result of meaningful learning in students. The maximum score of the questionnaire is 5. The scale is prepared to add the different items even if they measure different items. They will not be interpreted separately.
Learning behaviours (I) | 0, 4, 8, 12 and 20 weeks
  Number of downloads were retrieved and collected from the institution's Moodle platform Virtual ClassroomTM, through class progress
Learning behaviours (II) | 0, 4, 8, 12 and 20 weeks
  Number of topics visited were retrieved and collected from the institution's Moodle platform Virtual ClassroomTM, through class progress
Learning behaviours (III) | 0, 4, 8, 12 and 20 weeks
  The score of questionnaires were retrieved and collected from the institution's Moodle platform Virtual ClassroomTM, through class progress

CONTACTS AND LOCATIONS:
Overall Officials: David Hernández-Guillén, PT, PhD, Study Chair — University of Valencia
Locations (1):
- University of Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No